CLINICAL TRIAL: NCT06443827
Title: Effects of Intravenous Amantadine Sulphate on Brain Dynamics and Neurobehavioral Status in Patients With Disorders of Consciousness
Brief Title: Effect of Intravenous Amantadine Sulphate on Disorders of Consciousness
Acronym: DOC-AMSUL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Sanitaria dell'Alto Adige (Other)
Responsible Party: Principal Investigator, Viviana Versace, MD, Azienda Sanitaria dell'Alto Adige
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39049
Record Dates: First submitted 2024-05-15; First posted 2024-06-05 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Amantadine; Consciousness Disorders; Electroencephalography
Keywords: DoC = Disorders of Consciousness; PSD = Power Spectral Density; Amantadine sulphate; EEG
MeSH Terms: conditions — Consciousness Disorders | interventions — Amantadine

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover ("within subjects") study with an A-B-A-B treatment scheme, in which "placebo" (A) and "amantadine sulphate" (B) intervention sessions alternated weekly in the same patient for a total of four weeks (A1-B1-A2-B2).
Masking Description: Blindness about treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amantadine sulphate and placebo with schema A-B-A-B (Experimental): To obtain solid evidence of amantadine sulphate effects and their temporal dynamics, we conducted a double-blind, placebo-controlled, crossover ("within subjects") study with an A-B-A-B treatment scheme, in which "placebo" (A) and "amantadine sulphate" (B) intervention sessions alternated weekly in the same patient for a total of four weeks (A1-B1-A2-B2).
  Interventions: Drug: Amantadine Sulfate

INTERVENTIONS:
Drug: Amantadine Sulfate — intravenous amantadine sulphate at a single daily dose of 200 mg or physiological saline (0.9% NaCl solution)
  Other Names: physiological saline (0.9% NaCl solution)

SUMMARY:
Double-blind, placebo-controlled, crossover ("within subjects") study with an A-B-A-B treatment scheme to investigate the neuromodulatory effects of intravenous amantadine sulphate at a single daily dose of 200 mg in patients with disorders of consciousness (unresponsive wakefulness syndrome and minimally conscious state) by integrating traditional neurobehavioral assessment with spectral analysis of electrocortical activity derived from 64-channel electroencephalography (EEG) recordings.

DETAILED DESCRIPTION:
Research hypothesis Intravenous amantadine sulphate treatment (200 mg) over five days improves consciousness, defined as an increase in CRS-r score of at least 3 points, and changes the band powers of the EEG in patients with disorder of consciousness admitted in a Neurorehabilitation Department.

ELIGIBILITY:
Inclusion Criteria:

Adults with disorders of consciousness due to acquired brain injury classified according to international guidelines based on CRS-R evaluation as unresponsive wakefulness syndrome/vegetative state (UWS/VS) or minimally conscious state (MCS) either in the subacute or chronic stage

Exclusion Criteria:

* Age < 18 years
* History of epileptic seizures/status epilepticus
* Scalp defects
* pregnancy
* Severe uncompensated heart failure (NYHA IV)
* Atrioventricular block (AV block) second-degree and third-degree
* Known bradycardia (below 55 beats/minute)
* Known long QT interval (QTc according to Bazett > 420 ms
* History of serious ventricular arrhythmias
* Hypokalemia or hypomagnesemia
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) | days 14 and 28
  Increase in the Coma Recovery Scale-Revised (CRS-R) score of at least 1 point. The CRS-R consists of 23 items divided into six subscales designed to assess: Auditory (AU), Visual (V), Motor (M), Oromotor/Verbal (O), Communication (C), and Arousal functions (AR).
  The total score ranges between 0 (worst) and 23 (best). The subscales are composed of hierarchically ordered items; the lowest items (0) represent reflexive activity, while the highest items (4,5,6,3,2,3 points for AU, V, M, O, C respectively) represent cognitively mediated behaviours. We adopted a cut-off score of 8 for distinguish UWS/VS (<8) from MCS (≥8) in patients induced by amantadine sulphate vs. placebo
EEG band power alpha, beta, theta, delta | days 14 and 28
  Change in each canonical band power of EEG induced by amantadine sulphate

SECONDARY OUTCOMES:
"periodic" and "aperiodic" exponents of the average power spectral density | days 14 and 28
  Change in "periodic" and "aperiodic" exponents of the average power spectral density vs. placebo and vs healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Versace, MD, Principal Investigator — hospital of Vipiteno
Locations (1):
- Hospital of Vipiteno, Sterzing, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No